CLINICAL TRIAL: NCT06825156
Title: The Perioperative Renal and Metabolic Outcomes After Sodium Glucose Cotransporter 2 Inhibitor in Cardiac Surgery - an Open-label Phase IV Randomized Controlled Trial
Brief Title: Metabolic and Renal Outcomes in Cardiac Surgery Patients Receiving SGLT2 Inhibitors
Acronym: MERCURI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Lars Ivar Pieter Snel, Drs., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL78156.018.21
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Acute Kidney Injury
Keywords: CSA-AKI; SGLT-2i; Cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — empagliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: Single-center, open-label parallel-group randomized, controlled(usual care), phase IV clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Controlled (usual care) (No Intervention): Standard of care, Some additional blood drawn and urine collected to compare between both groups
- Intervention(Medication group) (Experimental): Patients receive 10mg Empagliflozin(SLGT-2i) daily from 3 days prior to surgery untill 2 days post-surgery which includes day of surgery.
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Patients receive 10mg Empagliflozin(SLGT-2i) daily from 3 days prior to surgery untill 2 days post-surgery which includes day of surgery.
  Other Names: Gliflozin; SGLT-2i
  Arms: Intervention(Medication group)

SUMMARY:
To investigate the potential of preoperative initiation (3 days) and perioperative continuation (until day 2 after surgery) of empagliflozin(sodium glucose co transporter 2 inhibitor(SGLT-2i)) 10 mg daily to reduce the acute kidney injury marker neutrophil gelatinase-associated lipocalin (NGAL) measured in serum and urine on day 2 postoperatively in patients undergoing cardiopulmonary bypass surgery by comparing a study medication group to a control group in an open-label set-up.

DETAILED DESCRIPTION:
Adult patients scheduled for elective cardiopulmonary bypass assisted cardiothoracic surgery will be informed about the study and after receiving informed consent will be divided between two groups in an openlabel fashion:

Intevention group: Takes study medication(10mg Empagliflozin once a day in the morning) 3 days prior to surgery, day of surgery and 2 days post-surgery.

Control group: follows the usual standard of care. At time moment before surgery and before medication is taken blood and urine sample is taken. This is repeated on day of surgery, and the consecutive 2 days after surgery.

Form these samples biomakers for kidney injury will be measured and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years old (inclusive)
* Undergoing elective cardiac surgery with cardio-pulmonary bypass.
* Providing informed consent

Exclusion Criteria:

Current treatment with SGLT2 inhibitors.

* Diabetes Mellitus Type 1
* BMI<25 for people with type 2 diabetes
* Reduced renal function at baseline with eGFR < 30 ml/min.
* Systolic blood pressure < 100 mmHg at time of inclusion.
* Emergency surgery, defined as in need of surgery for medical reasons < 7 days, i.e. "S1-4" according to the Amsterdam UMC classification.
* Female of child-bearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods.
* Known or suspected allergy to trial products or other drugs in the same class.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
NGAL | Day 2 post surgery
  Neutrophil gelatinase-associated lipocalin (NGAL) concentration in plasma on postoperative day 2

SECONDARY OUTCOMES:
Neutrophil gelatinase-associated lipocalin (NGAL) concentration in plasma. | Before surgery, day of surgery, day 1+2 after surgery
  NGAL measured in plasma
Kidney Injury Molecule-1 (KIM-1) in plasma. | Before surgery, day of surgery, day 1+2 after surgery
  KIM-1 concentration measured in plasma
Perioperative peak and average blood glucose levels, as measured during usual care. | During study per untill 4 days post-operatively
  Glucose levels recorded during usual routine care
Blood ketone levels. | During surgery at 4 measurement moments or during usual care.
  Blood ketones measured intra-operatively
Renal functioning (KDIGO criteria) | During study period untill post-operative day 4
  development of serum creatinine levels and urine output measured untill post-operative day 4

OTHER OUTCOMES:
Ketoacidosis | During study period untill post-operative day 4
  Incidence of keto-acidosis defined as combination of blood ketone concentration >3mmol/l in combination with high-anion gap acidosis ([Na+]-[Cl-]-[HCO3-]>12).
Hypoglycemia | During study period untill post-operative day 4
  Incidence of Hypoglycemia during study period

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hermanides, Dr., Principal Investigator — Amsterdam University Medical Centre
Locations (1):
- Amsterdam University Medical Centre, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Protocol
Supporting Information: Study Protocol, ICF
Time Frame: at least 5 years after publication
Access Criteria: Relevant reason to validate the request for access of this data

REFERENCES:
- See also: Link of the former published study protocol, National register of the Netherlands has ceased to exist. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2021-003172-13/NL